CLINICAL TRIAL: NCT01632150
Title: Phase 2a Single-Arm Safety Study of Elotuzumab in Combination With Thalidomide and Dexamethasone in Subjects With Relapsed and/or Refractory Multiple Myeloma
Brief Title: Safety Study of Elotuzumab in Combination With Thalidomide and Dexamethasone in Relapsed and/or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA204-010; 2011-005121-49 (EudraCT Number)
Record Dates: First submitted 2012-06-28; First posted 2012-07-02 (Estimated); Results first posted 2016-02-26 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-03

CONDITIONS: Relapsed and/or Refractory Multiple Myeloma
MeSH Terms: interventions — elotuzumab; Thalidomide; Dexamethasone; Calcium Dobesilate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Elotuzumab + Thalidomide + Dexamethasone + Cyclophosphamide (Experimental)
  Interventions: Biological: Elotuzumab; Biological: Thalidomide; Biological: Dexamethasone; Biological: Cyclophosphamide

INTERVENTIONS:
Biological: Elotuzumab — Powder for solution, 400-mg vials, for infusion
  Other Names: BMS-901608; HuLuc63
Biological: Thalidomide — 50-mg capsules administered orally
  Other Names: Thalomid®
Biological: Dexamethasone — 2- and 4-mg tablets (and various other strengths, as needed) administered orally and in 4- and 8-mg/mL (and various other strengths, as needed) solutions for intravenous administration
  Other Names: Decadron®; Dexamethasone Intensol®; Dexpak®; Taperpak®
Biological: Cyclophosphamide — 50-mg tablets administered orally
  Other Names: Cytoxan; Endoxan; Neosar

SUMMARY:
The purpose of this study is to determine the safety and tolerability of elotuzumab administered in combination with thalidomide and dexamethasone in the treatment of relapsed and/or refractory multiple myeloma.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Key Inclusion Criteria:

* Confirmed diagnosis of previously treated multiple myeloma with progression documented by criteria of the International Myeloma Working Group after or during the most recent therapy
* Patient received 5 or fewer prior lines of therapy
* Eastern Cooperative Oncology Group performance status of 0 or 1 (safety lead-in cohort) or 0 to 2 (additional patients)
* Measurable disease as defined by at least 1 of the following:

  * Serum immunoglobulin (Ig)G, IgA, IgM, or monoclonal (M) protein level ≥0.5 g/dL or serum IgD M protein level ≥0.05 g/dL; or
  * Urine M protein level ≥200 mg excreted in a 24-hour collection sample; or
  * Involved serum free light chain level ≥10 mg/dL, provided the free light chain ratio is abnormal

Key Exclusion Criteria:

* Solitary bone or solitary extramedullary plasmacytoma as the only evidence of plasma cell dyscrasia
* Monoclonal gammopathy of undetermined significance, smoldering myeloma, or Waldenström's macroglobulinemia
* Left ventricular ejection fraction by echocardiogram or Multi Gated Acquisition ≤50%
* Electrocardiogram finding of QTc ≥450 msec
* Active plasma cell leukemia (defined as either 20% of peripheral white blood cells, composed of plasma/CD138+ cells or an absolute plasma cell count of 2*10^9/L)
* Diagnosis of nonsecretory myeloma
* Active hepatitis A, B, or C virus infection
* Grade ≥2 neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-05; Primary Completion 2013-10 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (7):
- Spain (7):
  - Local Institution, Barcelona, Barcelona
  - Local Institution, Barcelona
  - Local Institution, LaLaguna, S Cruz Tener
  - Local Institution, Madrid
  - Local Institution, Salamanca
  - Local Institution, Seville
  - Local Institution, Zaragoza

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 51 participants enrolled, 40 received treatment. Of those 40, 11 had cyclophosphamide added to their regimens.
Groups:
- Thalidomide + Elotuzumab + Dexamethasone + Cyclophosphamide: Participants received thalidomide in 28-day cycles: 50 mg, for the first 2 weeks, escalated to 100 mg for the next 2 weeks and beginning with Cycle 2, to 200 mg once daily. Elotuzumab, 10 mg/kg, was administered as an intravenous infusion weekly for the first 2 cycles and beginning with Cycle 3, every 2 weeks. Dexamethasone, 40 mg, was administered weekly on those weeks when elotuzumab was not administered. On weeks when elotuzumab was also given, participants received dexamethasone as a split dose of 28 mg, 3 to 24 hours before the elotuzumab infusion, and 8 mg intravenously at least 45 minutes before the infusion. Those patients with suboptimal response, defined as evidence of progressive disease between end of Cycle 2 and end of Cycle 4 or inability to achieve partial response or better by end of Cycle 4, also received cyclophosphamide, 50 mg. Cyclophosphamide could not be added beyond Cycle 5.
Period: Overall Study
Arm/Group | Thalidomide + Elotuzumab + Dexamethasone + Cyclophosphamide
Started | 40
Received Cyclophosphamide | 11
Completed | 0 (Completed=still receiving treatment)
Not Completed | 40
Not completed — Disease progression | 27
Not completed — Study drug toxicity | 1
Not completed — Unrelated adverse event | 7
Not completed — Withdrawal by Subject | 2
Not completed — Patient underwent autologous transplant | 1
Not completed — Moved to compassionate program | 2

BASELINE CHARACTERISTICS:
Population: All participants who received thalidomide +elotuzumab + dexamethose (40) and had cyclophosphamide added to the regimen (11).
Arm/Group | Thalidomide + Elotuzumab + Dexamethasone + Cyclophosphamide
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.3 (8.47)
Age, Customized [Number; unit: Participants]
  Younger than 65 years | 22
  65 years and older to younger than 75 years | 12
  75 years and older | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 40
  More than one race | 0
  Unknown or Not Reported | 0
Myeloma type [Number; unit: Participants]
  Immunoglobulin (Ig)G | 15
  IGA | 7
  IGM | 0
  IGD | 0
  Light chain disease | 9
  Not reported | 9
Eastern Cooperative Oncology Group (ECOG) performance status [Number; unit: Participants] — ECOG is a 6-item scale used to assess disease progression, daily functioning, appropriate treatment, and prognosis. Performance status is scored on a scale ranging from 0-5, with (best score) 0=fully active and able to carry on all predisease performance without restriction and (worst score) 5=death.
  Participants
    Score 0 | 17
    Score 1 | 21
    Score 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Received Treatment Including Cyclophosphamide and Had Grade 3 or Higher Nonhematologic Adverse Events (AEs)
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=having certain, probable, possible, or unknown relationship to study drug. Grade (Gr) 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4=Life-threatening or disabling, Gr 5=Death.
Time Frame: From the first dose of study drug until the last dose of treatment, including cyclophosphamide treatment
Population: All participants who received thalidomide, elotuzumab, and dexamethasone (40) including those who had cyclophosphamide added to the regimen (11).
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Thalidomide + Elotuzumab + Dexamethasone + Cyclophosphamide
Number analyzed (Participants) | 40
Percentage of participants | 62.5 [NA to 72.9] — Only the upper bound of the CI was calculated

2. Secondary Outcome: Percentage of All Participants Who Received Treatment Including Cyclophosphamide and Had 1 Dose Reduction or Discontinued Due to an Adverse Event
Description: Elotuzumab dose reduction was not permitted. Thalidomide dose reduction, delay, interruptions, or discontinuation was permitted in the event of toxicity. Dexamethasone dose reduction was also permitted in the event of toxicity and in the setting of infusion reactions;dose delays were allowed as clinically indicated at the discretion of the investigator. Cyclophosphamide dose reduction, delay, interruption, or discontinuation was permitted in the event of toxicity.
Time Frame: From the first dose of study drug until the last dose of treatment, including cyclophosphamide treatment
Population: All participants who received thalidomide, elotuzumab, and dexamethasone (40), including those who had cyclophosphamide added to the regimen (11).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Thalidomide + Elotuzumab + Dexamethasone + Cyclophosphamide: Participants received thalidomide in 28-day cycles: 50 mg, for the first 2 weeks, escalated to 100 mg for the next 2 weeks, then beginning with Cycle 2, to 200 mg once daily. Elotuzumab, 10 mg/kg, was administered as an intravenous infusion weekly for the first 2 cycles, then beginning with Cycle 3, every 2 weeks. Dexamethasone, 40 mg, was administered weekly on those weeks when elotuzumab was not administered. On weeks when elotuzumab was also given, participants received dexamethasone as a split dose of 28 mg, 3 to 24 hours before the elotuzumab infusion, and 8 mg intravenously at least 45 minutes before the infusion. Those patients with suboptimal response, defined as evidence of progressive disease between end of Cycle 2 and end of Cycle 4 or inability to achieve partial response or better by end of Cycle 4, also received cyclophosphamide, 50 mg. Cyclophosphamide could not be added beyond Cycle 5.
Arm/Group | Thalidomide + Elotuzumab + Dexamethasone + Cyclophosphamide
Number analyzed (Participants) | 40
Percentage of participants | 65.0 [48.3 to 79.4]

3. Primary Outcome: Percentage of All Participants Who Received Treatment Without Cyclophosphamide and Had Grade 3 or Higher Nonhematologic Adverse Events (AEs)
Description: as for outcome 1
Time Frame: From the first dose of study drug until the earlier of discontinuation from E-Td or the time when cyclophosphamide was initiated
Population: All participants who received thalidomide + elotuzumab + dexamethasone regimen, from first dose of study drug until discontinuation or until cyclophosphamide was initiated, whichever came first.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Groups:
- Thalidomide + Elotuzumab + Dexamethasone: Participants received thalidomide in 28-day cycles: 50 mg, for the first 2 weeks, escalated to 100 mg for the next 2 weeks and beginning with Cycle 2, to 200 mg once daily. Elotuzumab, 10 mg/kg, was administered as an intravenous infusion weekly for the first 2 cycles, then beginning with Cycle 3, every 2 weeks. Dexamethasone, 40 mg, was administered weekly on those weeks when elotuzumab was not administered. On weeks when elotuzumab was also given, participants received dexamethasone as a split dose of 28 mg, 3 to 24 hours before the elotuzumab infusion, and 8 mg intravenously at least 45 minutes before the infusion.
Arm/Group | Thalidomide + Elotuzumab + Dexamethasone
Number analyzed (Participants) | 40
Percentage of participants | 55.0 [NA to 65.9] — Only the upper bound of the CI was calculated

4. Secondary Outcome: Percentage of All Participants Who Received Treatment Without Cyclophosphamide and Had 1 Dose Reduction or Discontinued Due to an Adverse Event
Description: Elotuzumab dose reduction was not permitted. Thalidomide dose reduction, delay, interruptions, or discontinuation was permitted in the event of toxicity. Dexamethasone dose reduction was also permitted in the event of toxicity and in the setting of infusion reactions;dose delays were allowed as clinically indicated at the discretion of the investigator.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Thalidomide + Elotuzumab + Dexamethasone: Participants received thalidomide in 28-day cycles: 50 mg, for the first 2 weeks, escalated to 100 mg for the next 2 weeks, then beginning with Cycle 2, to 200 mg once daily. Elotuzumab, 10 mg/kg, was administered as an intravenous infusion weekly for the first 2 cycles, then beginning with Cycle 3, every 2 weeks. Dexamethasone, 40 mg, was administered weekly on those weeks when elotuzumab was not administered. On weeks when elotuzumab was also given, participants received dexamethasone as a split dose of 28 mg, 3 to 24 hours before the elotuzumab infusion, and 8 mg intravenously at least 45 minutes before the infusion.
Arm/Group | Thalidomide + Elotuzumab + Dexamethasone
Number analyzed (Participants) | 40
Percentage of participants | 57.5 [40.9 to 73.0]

ADVERSE EVENTS:
Time Frame: From date of first dose to 60 days post last dose
Arm/Group | All Treated Subjects
Serious Adverse Events (participants affected / at risk) | 23/40
Other Adverse Events (participants affected / at risk) | 39/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Treated Subjects (N=40)
Cardio-respiratory arrest (Cardiac disorders) | 1
Myocarditis (Cardiac disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Cardiac death (General disorders) | 1
Disease progression (General disorders) | 1
Sudden death (General disorders) | 1
Aspergillus infection (Infections and infestations) | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 2
Lung infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Respiratory tract infection (Infections and infestations) | 4
Septic shock (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Aspiration bronchial (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Spinal cord compression (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Treated Subjects (N=40)
Anaemia (Blood and lymphatic system disorders) | 15
Neutropenia (Blood and lymphatic system disorders) | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 9
Diplopia (Eye disorders) | 2
Vision blurred (Eye disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 17
Chest pain (General disorders) | 2
Chills (General disorders) | 2
Crepitations (General disorders) | 2
Fatigue (General disorders) | 3
Gait disturbance (General disorders) | 2
Oedema peripheral (General disorders) | 12
Pain (General disorders) | 3
Pyrexia (General disorders) | 13
Gastroenteritis (Infections and infestations) | 2
Herpes zoster (Infections and infestations) | 3
Influenza (Infections and infestations) | 4
Lower respiratory tract infection (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 5
Respiratory tract infection (Infections and infestations) | 9
Upper respiratory tract infection (Infections and infestations) | 5
Blood creatinine increased (Investigations) | 3
Blood glucose increased (Investigations) | 2
Laboratory test abnormal (Investigations) | 2
Weight decreased (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 8
Iron deficiency (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 12
Bone pain (Musculoskeletal and connective tissue disorders) | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Dizziness (Nervous system disorders) | 7
Neuropathy peripheral (Nervous system disorders) | 11
Paraesthesia (Nervous system disorders) | 5
Somnolence (Nervous system disorders) | 4
Tremor (Nervous system disorders) | 5
Anxiety (Psychiatric disorders) | 5
Confusional state (Psychiatric disorders) | 2
Catarrh (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Deep vein thrombosis (Vascular disorders) | 4
Hypertension (Vascular disorders) | 4
Hypotension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.